CLINICAL TRIAL: NCT01310816
Title: A Phase 2, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of IPI-926 in Patients With Metastatic or Locally Advanced (Unresectable) Chondrosarcoma
Brief Title: A Safety and Efficacy Study of Patients With Metastatic or Locally Advanced (Unresectable) Chondrosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPI-926-04
Record Dates: First submitted 2011-03-03; First posted 2011-03-09 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Conventional Chondrosarcoma
Keywords: malignant neoplasms of the bone; bone sarcoma
MeSH Terms: conditions — Bone Neoplasms | interventions — IPI-926

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPI-926 (Active Comparator): IPI-926
  Interventions: Drug: IPI-926
- Sugar Pill (Placebo Comparator): Placebo Arm, sugar pill
  Interventions: Drug: Placebo Arm

INTERVENTIONS:
Drug: IPI-926 — Oral
  Arms: IPI-926
Drug: Placebo Arm — oral placebo
  Arms: Sugar Pill

SUMMARY:
IPI-926 is an inhibitor of the hedgehog pathway. IPI-926 may improve therapeutic outcomes in patients with Chondrosarcoma.

DETAILED DESCRIPTION:
Study IPI-926-04 is a Phase 2, double-blind, placebo-controlled, multicenter, trial evaluating the safety and efficacy of IPI-926 in patients with metastatic or locally advanced (unresectable) chondrosarcoma. The study includes an optional cross-over to open-label IPI-926 for patients randomly assigned to placebo who experience documented disease progression.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing informed consent.
* Pathologically diagnosed conventional chondrosarcoma. Patients must have tumor sample(s) available or provide tumor samples from a new biopsy
* Metastasis to at least 1 location or locally advanced disease that is deemed unresectable by a surgeon
* At least 1 radiologically measurable target lesion per RECIST 1.1.
* Patients must have documented radiographic progression of disease within the 6-month period prior to screening. (MRI or CT Scan)
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1.
* Life expectancy of at least 3 months
* All women of child-bearing potential (WCBP), all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study and for 30 days after the last dose of study drug.
* Ability to adhere to the study visit schedule and all protocol requirements.
* Voluntarily signed an informed consent form.

Exclusion Criteria:

* Other invasive malignancies diagnosed within the last 5 years, except non-melanoma skin cancer and localized cured prostate and cervical cancer.
* Systemic anti-cancer therapy within 21 days prior to the first dose of study drug, or radiotherapy within 14 days prior to the first dose of study drug.
* Prior treatment with a Hedgehog pathway inhibitor
* Medically significant surgical procedures or significant traumatic injury within 28 days before Day 1.
* Inadequate hematologic function defined by:
* Hemoglobin <8.0 g/dL (80 g/L) (may be increased to this level with transfusion as long as there is no evidence of active bleeding).
* Inadequate hepatic function defined by:
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN).
* Total bilirubin >1.5 x ULN (with the exception of patients with Gilbert's disease).
* Cirrhotic liver disease, ongoing alcohol abuse, or known chronic active or acute hepatitis.
* Inadequate renal function defined by serum creatinine >1.5 x ULN
* Patients with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
* Presence of active infection or systemic use of antibiotics within 72 hours of treatment.
* Significant co-morbid condition or disease, which in the judgment of the Investigator, would place the patient at undue risk or interfere with the study. Examples include, but are not limited to sepsis and recent significant traumatic injury.
* Known human immunodeficiency virus (HIV) positivity.
* Known hypersensitivity to IPI-926, or any of the excipients in IPI-926 or placebo capsules.
* Pregnant or lactating women.
* Current administration of the medications or foods which are known to be moderate or strong inhibitors of CYP3A4 activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | estimated 6 months
  * To compare progression-free survival (PFS) in patients with metastatic or locally advanced (unresectable) chondrosarcoma administered IPI-926 or placebo.
  * Number of Incidence of reported adverse events and abnormal laboratory test results. To evaluate the safety of IPI-926 or placebo in patients with metastatic or locally advanced (unresectable) chondrosarcoma

SECONDARY OUTCOMES:
Comparison of Time To Progression (TTP) | estimated 6 months
  *To compare, Time To Progression (TTP) with metastatic or locally advanced (unresectable) chondrosarcoma patients administered IPI-926 or placebo
Comparison of Overall Survival (OS) | estimated 6 months
  To compare Overall Survival (OS) with metastatic or locally advanced (unresectable) chondrosarcoma patients administered IPI-926 or placebo
Overall Response Rate (ORR) | estimated 6 months
  To compare Overall Response Rate (ORR) with metastatic or locally advanced (unresectable) chondrosarcoma patients administered IPI-926 or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Santabarbara, MD, Study Chair — Infinity Pharmaceuticals, Inc.
Locations (36):
- United States (15):
  - (TGen) Translational Genomics Research Institute, Scottsdale, Arizona
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - Sydney Cancer Centre, Camperdown, New South Wales
  - Monash Medical Centre, East Bentleigh, Victoria
- Medizinische Universität Wien, Vienna, Vienna, Austria
- Mount Sinai Hospital, Toronto, Ontario, Canada
- France (3):
  - Centre Léon Bérard, Service d'Oncologie Médicale, Lyon, Auvergne-Rhône-Alpes
  - Centre René Gauducheau, Saint-Herblain, Pays de la Loire Region
  - Institut de Cancérologie Gustave Roussy, Villejuif, Île-de-France Region
- Germany (3):
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Helios Klinikum Bad Saarow, Bad Saarow, Brandenburg
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
- Italy (2):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano
- Leids Unversitair Medisch Centrum, Leiden, South Holland, Netherlands
- Radiumhospitalet, Oslo, Norway
- Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie w Warszawie, Warsaw, Masovian Voivodeship, Poland
- Russia (2):
  - SI Russian Oncological Research Center, Moscow, Moscow
  - Moscow n.a. P.A Herzen Oncology Research Institute of Rosmedtechnologies, Moscow, Moscow
- Skånes Universitetssjukhus, Lund, Skåne County, Sweden
- United Kingdom (3):
  - Royal Orthopaedic Hospital, Birmingham, England
  - University College Hospital, London, England
  - Newcastle General Hospital, Newcastle upon Tyne, England